CLINICAL TRIAL: NCT03380754
Title: Effects of Preoperative Carbohydrate Rich Drinks on Immediate Postoperative Outcome in Total Knee Arthroplasty
Acronym: PONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Michael Charters, MD, Principal Investigator, MD, Adult Joint Reconstruction, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11180
Record Dates: First submitted 2017-10-31; First posted 2017-12-21 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Post Operative Nausea and Vomiting
Keywords: Nausea; Vomiting; Knee Arthroplasty; PONV; TKA
MeSH Terms: conditions — Vomiting; Nausea; Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blinded, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Research assistant who is not involved in any of the patients clinical care is responsible for randomization collection of data. All others are blinded to the groups involved.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Carbohydrate Rich Drink (Experimental): Group A will receive the carbohydrate rich drink, Nutricia preOp. This is the intervention group.
  Interventions: Dietary Supplement: Nutricia preOp
- Placebo Drink (Placebo Comparator): Group B will receive placebo, Nestle Splash Lemon Flavor Water (Placebo) (similarly flavored and appearing water, however with no calorie, carbohydrate or nutritional content).
  Interventions: Other: Nestle Splash Lemon Flavor Water (Placebo)
- No Drink (No Intervention): Group C will not receive any drink. This group will follow normal protocol.

INTERVENTIONS:
Dietary Supplement: Nutricia preOp — A clear, non-carbonated lemon-flavored, iso-osmolar carbohydrate drink for preoperative surgical patients. Used in studies supporting the Enhanced Recovery After Surgery (ERAS) Society Consensus Guidelines.
  Other Names: Carbohydrate rich drink
  Arms: Carbohydrate Rich Drink
Other: Nestle Splash Lemon Flavor Water (Placebo) — Placebo control drink. PURIFIED WATER, NATURAL FLAVORS, CITRIC ACID, SODIUM POLYPHOSPHATE, POTASSIUM SORBATE (PRESERVE FRESHNESS), POTASSIUM BENZOATE (PRESERVE FRESHNESS), SUCRALOSE, ACESULFAME POTASSIUM, CALCIUM DISODIUM EDTA, MAGNESIUM SULFATE.
  Arms: Placebo Drink

SUMMARY:
The aim of this study is to investigate the effect of preoperative carbohydrate rich drinks on postoperative nausea and vomiting in total knee arthroplasty. This is a prospective, double blinded, randomized controlled trial.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) continues to pose serious challenge to orthopaedic adult reconstructive surgeons, even after recent advances in anesthesia and improvements in perioperative care. Preoperative carbohydrate loading has been well studied in non-arthroplasty surgical fields. It has been shown to benefits which include decreased postoperative catabolism and insulin resistance, dampened metabolic stress response, thus decreased postoperative pain, anxiety, nausea, and vomiting. To the investigators knowledge, there is currently no literature describing the effects of preoperative carbohydrate rich drinks (CHO) in the setting of elective total joint arthroplasty. Using a prospective, randomized, double blind, placebo controlled model, the investigators aim to determine the effect of CHO on PONV in total knee arthroplasty.

The investigators plan to include a total of 150 patients in this study. All the arthroplasty surgeons at HF Main Campus expect to participate. Estimating approximately 20 patients enrolled per month, enrollment would likely occur over time span of 8 months.

Patients who are scheduled for elective, primary total knee arthroplasty will be recruited and consented in preoperative clinic visit according to the inclusion and exclusion criteria as outlined. Screening and consenting will be performed by the orthopaedic surgeon, resident, physician assistant, or nurse practitioner in clinic, who will be trained for this study. Patients who elect to participate will be randomized to CHO drink (Group A), placebo drink (Group B), or traditional fasting/no drink (Group C). Randomization will occur prior to enrollment in batches of twenty. Patients and treatment team will be blinded to the assignment. Enrolled subjects will be given a kit which will include study information, instructions for participation, data collection questionnaire (included with this submission), multiple-alarm timer, and two beverage bottles (labeled Drink 1 and Drink 2) for those in Group A or B. Group C will receive the kit, but without beverage. A research assistant who is not involved in any of the subjects' care will be responsible for preparation of the kits.

Beverage in Group A will consist of a clear, non-carbonated lemon-flavored, iso-osmolar carbohydrate drink (Nutricia preOp; 12.5% carbohydrates, 50kcal/100mL, 260mOsm/kg, pH 5.0). This drink has been previously used in studies supporting Enhanced Recovery After Surgery (ERAS) Society Consensus Guidelines. Beverage in Group B will consist of the same quantity of clear, lemon flavored water (Nestle Splash Lemon; 0kcal/100mL). All beverages will be bottled in clear PET plastic IPEC tamper evident bottles. Bottles will be labeled Drink 1 (800 mL) or Drink 2 (400 mL). Neither subjects nor treatment team will be able to identify type of beverage, however each drink label will include a special code, available only to research assistant to be able to identify contents of bottle (treatment vs placebo).

During the evening before surgery (8:00-10:00 PM), subjects in Group A and B will consume Drink 1 (800 mL) of their respective drink. After midnight, nothing will be allowed by mouth, except for except for single morning dose of appropriate drink (Drink 2, 400 mL) in Group A and Group B. Subjects will be instructed to consume morning drink 3 hours prior to scheduled time of surgery, and be completely consumed at least 2 hours prior to surgery.

Remainder of perioperative care will be standardized and occur according to routine care for Henry Ford Joints Protocol. Henry Ford Main Campus Perioperative Primary Total Joints Protocol is included with this submission for reference. All patients will receive epidural for anesthesia. All patients will receive dexamethasone 10mg IV x 1 dose preoperatively. All patients will have ondansetron 4mg IV Q6 hours as needed available postoperatively. Multimodal perioperative pain management regimen will be standardize according to protocol.

Postoperatively, data points will be recorded by nurse in electronic medical record: events of nausea and vomiting, medication consumption, and pain VAS scores. These data points will be collected and separated by postop 0-4 hours, 4-12 hours, and 12-24 hours. Additionally, subjects will be reminded to fill out their questionnaire in preop, 4 hours postop, 12 hours postop, and 24 hours postop (questionnaire is included in this submission). Primary goal is to compare incidence and timing of postoperative nausea and vomiting between groups.

The drink/placebo will be supplied to the patient by the treating surgeon, physician assistant, or orthopaedic resident in clinic at the time of the last preoperative clinic visit prior to surgery. The appropriate drink will be included in a "kit" that will be given to the patient at that time. The kit will include study information, instructions for participation, the data collection questionnaire (included with this submission), a multiple-alarm timer, and two beverage bottles (labeled Drink 1 and Drink 2) for those in Group A or B. Group C will receive the same kit with all the same contents, but without a beverage.

The drinks will be mixed and bottled by the research assistant, and will be "ready to drink" upon receipt by the participant. This will be performed in batches of 20 to prevent any shelf-life errors. The carbohydrate rich drink (Nutricia preOp) is purchased in powder form with included instructions on mixing. Each patient package comes with 6 powder packs. The powder will be mixed in appropriate plastic beverage container with purified drinking water. Purified water will be room temperature at time of mixing, per Nutricia instructions. Drinks will be mixed in their respective beverage container according to manufacturer instruction: Drink 1 is 800 cc (4 powder packs), and drink 2 is 400 cc (2 powder packs). This drink will therefore appear clear and similar to the placebo group. For the placebo group, the appropriate amount of Nestle Splash Lemon flavored water will be poured into the appropriate bottles. Bottles will be capped with tamper evident caps. "Ready to drink" beverages will then be included in the appropriate kits by the research assistant. The kits will then be stored in a cool place, locked, away from light, in one of the K12 clinic offices. All mixing and bottling will be performed with use of standard sanitary precautions by one person, the research assistant. The research assistant will also be responsible for labelling and coding the drinks to allow for identification of the drinks.

The questionnaire will be included in the kit, which is given to the patient at their last preoperative visit prior to surgery. The kit will also include a handheld multiple-alarm timing device, which will be used to ensure patients complete the appropriate sections of their questionnaire at the requested time points. In the preoperative holding area, the patients will simply be reminded by the staff, resident, or surgeon, to complete the "preop" portion of the questionnaire. Post-operatively, the multiple-alarm timer will be utilized to standardize timing of responses. The timer will be programmed appropriately before surgery, and will be "started" by the orthopaedic resident postoperatively once the patient is dropped off in the recovery unit following surgery. The handheld timer will be pre-programmed to sound an alarm at time points 4 hours, 12 hours, and 24 hours post surgery.

Patients themselves will be mostly responsible for ensuring they comply with the requested time points in completing the questionnaire. However, the orthopaedic floor nurses will also be educated on this study and will encourage/assist in administration of the questionnaire when needed. The nurse will collect the questionnaire once it is complete, prior to patient discharge. The nursing station will have a specific folder where each questionnaire will be placed following completion. The research assistant will check folder daily, and items will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years of age) scheduled for elective, unilateral, primary total knee arthroplasty
* Able to give valid consent

Exclusion Criteria:

* Impaired gastrointestinal motility
* On pro-motility medication
* Pregnancy
* HbA1c > 7.5
* Fasting glucose >200
* Acquired immunodeficiency
* Renal failure (creatinine > 2 mg/dL)
* Cirrhosis
* Severe malnutrition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Post operative nausea | 4 hours postoperatively
  Nausea, assess by questionnaire, 10 point scale (0 = no nausea, 10 = very nauseous, and medical record.
Post operative nausea | 12 hours postoperatively
  Nausea, assess by questionnaire, 10 point scale (0 = no nausea, 10 = very nauseous, and medical record.
Post operative nausea | 24 hours postoperatively
  Nausea, assess by questionnaire, 10 point scale (0 = no nausea, 10 = very nauseous, and medical record.
Post operative vomiting | 4 hours postoperatively
  Vomiting, assess by questionnaire, 10 point scale (0 = no vomiting, 10 = copious emesis, and medical record notes of emesis.
Post operative vomiting | 12 hours postoperatively
  Vomiting, assess by questionnaire, 10 point scale (0 = no vomiting, 10 = copious emesis, and medical record notes of emesis.
Post operative vomiting | 24 hours postoperatively
  Vomiting, assess by questionnaire, 10 point scale (0 = no vomiting, 10 = copious emesis, and medical record notes of emesis.

SECONDARY OUTCOMES:
Length of hospital stay | From the time of hospital admission following surgery, until the time of hospital discharge as recorded in EMR, assessed up to 1 month
  Length of stay recorded in hours
Post operative opiate consumption | From the time of surgery until the time of hospital discharge, assessed up to 72 hours postoperatively
  Morphine equivalents, opiates assessed by medical record
Post operative pain scores | From the time of surgery until the time of hospital discharge, assessed up to 72 hours postoperatively
  Pain, 10 point visual analog pain scale (0 = no pain, 10 = worst pain ever)
Peri operative hunger and discomfort | 4 hours, 12 hours, and 24 hours postoperatively
  Hunger and discomfort, 10 point hunger scale (0 = satiated and comfortable, 10 = very hungry and uncomfortable)
Incidence of secondary adverse events | From the time of surgery until the time of hospital discharge, assessed up to 1 month postoperatively
  pulmonary aspiration, delay of surgery due to consumption of drink.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Charters, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
There are currently no plans to share participant data with other researchers.

REFERENCES:
- [Derived] Kadado A, Shaw JH, Ayoola AS, Akioyamen NO, North WT, Charters MA. Effects of Preoperative Carbohydrate-rich Drinks on Immediate Postoperative Outcomes in Total Knee Arthroplasty: A Randomized Controlled Trial. J Am Acad Orthop Surg. 2022 Jun 1;30(11):e833-e841. doi: 10.5435/JAAOS-D-21-00960. Epub 2022 Mar 18. PMID 35312650